CLINICAL TRIAL: NCT01993797
Title: Lung Ultrasound: a Useful Tool in Diagnosis and Management of Bronchiolitis?
Brief Title: Lung Ultrasound in Diagnosis and Management of Bronchiolitis Bronchiolitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: S. Giacomo Hospital (Other)
Collaborators: University of Bari (Other)
Responsible Party: Principal Investigator, Mariano Manzionna, Director of Pediatric Unit, S. Giacomo Hospital
Other Study IDs: MMSGH
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bronchiolitis: children presented with signs suggestive of bronchiolitis
  Interventions: Other: Lung US

INTERVENTIONS:
Other: Lung US

SUMMARY:
To evaluate the correlation between clinical and ultrasound findings in children presented with signs suggestive of bronchiolitis and to validate an ultrasound score for bronchiolitis that will correlate with specific clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* children presented with signs suggestive of bronchiolitis

Exclusion Criteria:

* other major pathology

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children presented with signs suggestive of bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
clinical and ultrasound findings | baseline
  To evaluate the correlation between clinical and ultrasound findings in children presented with signs suggestive of bronchiolitis

SECONDARY OUTCOMES:
ultrasound score for bronchiolitis and clinical outcome | baseline
  to validate an ultrasound score for bronchiolitis that will correlate with specific clinical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- S Giacomo Hospital, Monopoli, Bari, Italy

REFERENCES:
- [Background] Caiulo VA, Gargani L, Caiulo S, Fisicaro A, Moramarco F, Latini G, Picano E. Lung ultrasound in bronchiolitis: comparison with chest X-ray. Eur J Pediatr. 2011 Nov;170(11):1427-33. doi: 10.1007/s00431-011-1461-2. Epub 2011 Apr 6. PMID 21468639
- [Derived] Basile V, Di Mauro A, Scalini E, Comes P, Lofu I, Mostert M, Tafuri S, Manzionna MM. Lung ultrasound: a useful tool in diagnosis and management of bronchiolitis. BMC Pediatr. 2015 May 21;15:63. doi: 10.1186/s12887-015-0380-1. PMID 25993984